### Republic of Turkey

### **Black Sea Technical University Rectorate**

### **Directorate of the Institute of Health Sciences**

**Number:** 27863166-302.14.04- 02/22/2024 22.02.2024 22.02.2024

**Subject:** Thesis Proposal (Berrin GÖGER)

### TO THE DEPARTMENT OF NURSING

Regarding the "Doctoral Thesis Proposal" of Berrin GÖGER, a doctoral student in your department, a copy of the Institute Management Board decision dated 14.02.2024 and numbered 160 is attached. I kindly request your attention and action.

Assistant Professor Efnan ABDIOĞLU FAZLI

Director a.

Deputy Director of the Institute

## DATA COLLECTION TOOLS

Newborn Baby Identification Information Form

Baby Group No:

| Date: / |
|---|
| 1. Gender: ( ) Female ( ) Male |
| 2. Gestational Age (specify in weeks): |
| 3. Mode of Delivery: |
| 4. Birth Weight |
| 5. Birth Length: |
| 6. Postnatal Age (specify in days): |
| 7. Current Weight: |
| 8. Current Height: |
| 9. Baby's feeding method: ( ) Breast milk ( ) Formula ( ) Breast milk + formula |

# **Parent Information Form**

Parent Group No: Date: / /

| 1. Mother's age: |
|---|
| 2. Mother's education level: ( ) Illiterate ( ) Primary school ( ) Middle school ( ) High school ( ) College and above |
| 3. Mother's occupation: ( ) Not working ( ) Civil servant ( ) Worker ( ) Self-employed ( ) Retired |
| 4. Father's age: |
| 5. Father's education level: ( ) Illiterate ( ) Primary school ( ) Middle school ( ) High school ( ) University and above |
| 6. Father's occupation: ( ) Not working ( ) Civil servant ( ) Worker ( ) Self-employed ( ) Retired |

### **Newborn Baby Observation Form**

Baby Group No: Date: / /

### Crying duration:

Baby's body temperature before the procedure:

Baby's body temperature after the procedure:

Baby's respiratory rate before the procedure:

Baby's respiratory rate after the procedure:

### PHYSIOLOGICAL PARAMETERS

1 MINUTE BEFORE THE PROCEDURE
DURING THE PROCEDURE
1 MINUTE AFTER THE PROCEDURE
OXYGEN SATURATION
HEART RATE

#### **Neonatal Infant Pain Scale (NIPS)**

Infant Group No.:
Date: / /

### Categories 0 1 2

Facial expression Calm face, natural expression Tense facial muscles, wrinkled forehead and chin

Crying Silent, not crying Mild whimpering, intermittent crying Screaming, wailing, loud, continuous crying

Breathing pattern Normal breathing Variable, irregular, faster than normal breathing, gasping

Arms No muscle rigidity, often random arm movements Tense, straight arms, stiff and/or rapid extension/flexion

Legs No muscle rigidity, often random leg movements Tense, straight legs, stiff and/or rapid extension/flexion

State of alertness Quiet, peaceful, sleeping and/or calm Lively, restless, and unable to be calmed

### **Voluntary Consent Form**

Dear Parent,

You and Your Baby

You are participating in a scientific study titled "The Effect of Mechanical Vibration and Tapping Methods on Reducing Pain During Hepatitis B Vaccination in Infants."

Your participation in this study is voluntary. By checking the consent box below, you will be able to begin answering the questionnaire, and data will be collected from your baby using data collection tools before, during, and after the procedure, without any intervention such as mechanical vibration or tapping.

Your honest answers to the survey questions are crucial for the study to yield accurate results. The answers you provide will be used for scientific purposes, kept strictly confidential, and will not be shared with others.

Thank you.

Lecturer Berrin GÖGER

☐ I agree to participate in the study voluntarily.